CLINICAL TRIAL: NCT01464502
Title: A Prospective Randomised Controlled Trial of Cardiac Resynchronisation Therapy Guided by Invasive dP/dT: Radi-CRT Study
Brief Title: Pressure Wire Guided Cardiac Resynchronisation Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Manav Sohal, Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/LO/1879
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac resynchronisation therapy; Acute haemodynamic response; Responder
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard CRT Implant (Active Comparator)
  Interventions: Procedure: Standard CRT Implant
- Pressure-wire guided CRT Implant (Active Comparator)
  Interventions: Procedure: Pressure-wire guided CRT implant

INTERVENTIONS:
Procedure: Standard CRT Implant
  Arms: Standard CRT Implant
Procedure: Pressure-wire guided CRT implant — A pressure wire will be sited in the left ventricle to measure dP/dT max. The LV lead position that gives the highest dP/dT max will be the final position used.
  Arms: Pressure-wire guided CRT Implant

SUMMARY:
Heart failure patients may benefit from having a special pacemaker implanted that can make the heart pump in a more coordinated and efficient way Cardiac Resynchronisation Therapy (CRT). For the heart to pump well it is necessary for the pacing wires to be placed in optimal positions. Only two thirds of people respond to CRT and this may be because of non-ideal pacing wire position. A potential marker for response is the change in heart pump pressure change over time. The aim of this study is to use a specialised wire in the main pumping chamber of the heart to record the pressure changes with the pacing lead in various positions to determine the optimal position. It is postulated that the improved pressure changes will increase the proportion of responders.

Pilot study work has shown that the work is technically feasible and safe. The initial data has been published in a highly regarded scientific journal. This main study will be a multicentre randomised controlled trial whereby patients will be randomised to either standard treatment or pressure wireguided treatment. The patients in the pressurewire guided arm will have a specialised wire implanted into the main pumping chamber of their heart via a blood vessel at the top of the leg (or less commonly a blood vessel in the wrist). This will measure acute pressure changes over time and the pacing lead will be positioned in the site that gives the greatest change in pressure.

If the patients in the pressurewire guided arm fare better than those receiving standard treatment it may alter how a large proportion of heart failure patients are treated around the world. The study requires 282 patients and is likely to take two years to complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling standard criteria for CRT
* Ischaemic or non-ischaemic heart failure

Exclusion Criteria:

* Contraindication to pressure wire assessment including:
* Severe aortic valve disease
* Mechanical aortic valve replacement
* Severe peripheral vascular disease
* LV thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion of CRT responders at 6 months | 6 months
Change in clinical composite score at 6 months | 6 months

SECONDARY OUTCOMES:
Change in echo derived endsystolic volume (ESV) at six months | 6 months
Change in echo derived enddiastolic colume (EDV) at six months | 6 months
Change in echo derived left ventricular ejection fraction (LVEF) at 6 months | 6 months
Six month assessment of change in symptoms (Minnesota Living with Heart Failure Questionnaire) | 6 months
Six month change in 6 minute walk distance | 6 months
Six month change in VO2 max (CPET) | 6 months
Six month change in ntProBNP | 6 months
Six month difference in hospital readmission (days) | 6 months
Six month difference in mortality | 6 months
Difference in rates of successful LV lead implantation | One week
Difference in procedure duration | One week
Difference in radiation dose | One week
Difference in contrast dose | One week
Procedural complications | 6 months

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (2):
  - Hospital Auxolgico, Milan
  - San Rafaelle Hospital, Milan
- United Kingdom (8):
  - Medway Maritime Hospital, Gillingham, Kent
  - Guy's and St. Thomas' NHS Foundation NHS Trust, London, London
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Queen Elizabeth Hospital Woolwich, London
  - The Heart Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford